CLINICAL TRIAL: NCT03316313
Title: Prospective Cohort Study: Hepatitis C Screening in the Primary Care Setting
Brief Title: Hepatitis C Screening in the Primary Care Setting
Status: Completed | Type: Observational
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: BHS-1194
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C
Keywords: Public Health; Patient Education as Topic; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Date of birth: Those people born within the years 1945-1965
  Interventions: Diagnostic Test: Hepatitis C Antibody

INTERVENTIONS:
Diagnostic Test: Hepatitis C Antibody — Patients who received a blood test to screen for the Hepatitis C virus.

SUMMARY:
The purpose of this study is to determine whether patient education improves Hepatitis C screening in the primary care setting.

DETAILED DESCRIPTION:
Hepatitis C is a chronic, asymptomatic infection that progresses to liver cirrhosis and cancer in the later stages if left untreated. The Centers for Disease Control (CDC) recommends a one-time screening for high risk birth cohort between the years 1945-1965. Prior studies have evaluated methods to improve screening for hepatitis c with focus on increasing awareness in health professionals. Targets included nursing staff and electronic medical records. This study targets providing patients with education resources to see if screening rates improve.

ELIGIBILITY:
Inclusion Criteria:

* All patients born between the years 1945 and 1965.

Exclusion Criteria:

* Patients who had already received a prior screening test for Hepatitis C before the office visit.

Ages: 50 Years to 71 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Screening was performed at two locations with differing socioeconomic data per census reports.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of Patients Screened for Hepatitis C | June 2016 to October 2016.
  Change from baseline in number of patients from high-risk birth cohort screened for Hepatitis C during intervention period.

IPD SHARING:
Plan to Share IPD: No